CLINICAL TRIAL: NCT04877678
Title: Effects of Second-generation Antihistamine Bepotastine on Cough Outcomes in Cough Patients With Allergic Rhinitis: A Randomized, Double-blind, Placebo Controlled Study
Brief Title: Effects of Second-generation Antihistamine Bepotastine on Cough Outcomes in Cough Patients With Allergic Rhinitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Woo-Jung Song, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2021-0363
Record Dates: First submitted 2021-05-04; First posted 2021-05-07 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2023-01

CONDITIONS: Allergic Rhinitis; Cough
Keywords: cough, allergic rhinitis, antihistamines
MeSH Terms: conditions — Rhinitis, Allergic; Cough | interventions — bepotastine

STUDY DESIGN:
Intervention Model Description: A Randomized, Double-blind, Placebo Controlled Study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Allocation of medication is conducted by an independent physician who is not a co-investigator of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment group (Active Comparator): Participants will be treated with bepotastine.
  Interventions: Drug: Bepotastine
- Placebo group (Placebo Comparator): Participants will be treated with identical looking placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bepotastine — 10 mg Bepotastine, twice a day
  Other Names: Beposta B
  Arms: Treatment group
Drug: Placebo — Identical looking placebo, twice a day
  Arms: Placebo group

SUMMARY:
This is a phase 4 study to evaluate the the efficacy of second generation antihistamine on cough outcomes in cough patients with allergic rhinitis.

DETAILED DESCRIPTION:
This is a randomized, double blind, placebo controlled trial in which a total of 78 participants who have cough (≥ 3 weeks) and symptoms of allergic rhinitis will be enrolled. Study participants will be randomly assigned to either active treatment or placebo group. The subjects in active treatment groups will be treated with daily oral bepotastine for 2 weeks, while those in placebo group will take identical-looking tablets. The efficacy of bepotastine will be assessed at the end of 2-week intervention using leicester cough questionnaire.

ELIGIBILITY:
Inclusion Criteria:

1. Had a cough for at least 3 weeks (score of ≥30 mm on the VAS)
2. History or allergic rhinitis confirmed with skin prick test or serum specific IgE test AND current one or more symptoms of allergic rhinitis (runny nose, obstruction, sneezing, nasal itching)
3. Provided written informed consent
4. Were willing and able to comply with the study protocol

Exclusion Criteria:

1. Current smoker or individuals who have smoked within the past 1 month prior to study entry
2. Sings of coexisting respiratory diseases requiring active treatment such as fever, chills, wheezing, dyspnea, or purulent sputum
3. Currently under allergen immunotherapy
4. 1) Allergic rhinitis or chronic rhinosinusitis under treatment with intranasal corticosteroids (INS) or leukotriene receptor antagonist (LTRA) or 2) allergic rhinitis requiring treatment with INS or LTRA
5. Treatment with an angiotensin converting enzyme (ACE)-inhibitor within 4 weeks prior to the enrollment
6. Forced Expiratory Volume in 1 second (FEV1)/Forced Vital Capacity (FVC) < 0.7 or FEV1 % of predicted < 80% within 1 month prior to enrollment
7. Abnormal findings on chest x-ray related to cough within 1 month prior to enrollment
8. Diagnosis or treatment of bronchial asthma or COPD within 1 year of the enrollment
9. Clinically significant medical conditions possibly affecting evaluation of cough and nasal symptoms
10. History of hypersensitivity or severe adverse reaction to antihistamines
11. Unable to fill in the questionnaires (blindness, unable to read)
12. Unable to provide informed consent
13. History of taking following medication within 2 weeks of the enrollment; LTRA, nasal decongestants, intranasal corticosteroids (INS), systemic corticosteroids, antitussive agents (OTCs, codeine)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Leicester Cough Questionnaire (LCQ) | At baseline, and at 2 weeks of treatment
  The total score range of Leicester Cough Questionnaire is from 3 to 21. A higher score indicates a better quality of life.

SECONDARY OUTCOMES:
Visual analogue scale (VAS) of cough | At baseline, and at 2 weeks of treatment
  The visual analogue scale of cough ranges from 0-100. A higher score indicates more severe cough.
Cough hypersensitivity questionnaire (CHQ) | At baseline, and at 2 weeks of treatment
  The total score of cough hypersensitivity questionnaire ranges from 0-23. A higher score indicates a greater number of sensations or triggers associated with cough (or a higher degree of cough hypersensitivity).
Sino-nasal outcome test -22 (SNOT-22) | At baseline, and at 2 weeks of treatment
  The total score of sino-nasal outcome test -22 ranges from 0-110. A higher score indicates worse quality of life related to nasal symptoms.
Visual analogue scale (VAS) of globus pharyngeus | At baseline, and at 2 weeks of treatment
  The visual analogue scale of globus pharyngeus ranges from 0-100. A higher score indicates more severe sensation of globus pharyngeus.
Daily cough severity | daily assessment
  The scale of daily cough severity ranges from 0-10. A higher score indicates more severe cough.
Rate of adverse events | during 2 weeks of treatment
  Rate of adverse events in participant
Objective cough frequency | At baseline, and at 2 weeks of treatment
  24-hour objective cough frequency will be measured using the Hyfe Cough Tracker, a smartphone application-based cough monitoring. The measurement is optional and will be done in patients who agree to measure it.

CONTACTS AND LOCATIONS:
Overall Officials: Woo-Jung Song, Principal Investigator — Asan Medical Center
Locations (1):
- Asan medical center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No